CLINICAL TRIAL: NCT06518564
Title: A Phase 2 Study of Avelumab in Combination With ATR Inhibitor M1774 in Patients With ARID1A-mutated Recurrent Endometrial Cancer Who Have Received Prior Immunotherapy
Brief Title: Avelumab and M1774 in ARID1A-mutated Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Panagiotis Konstantinopoulos, MD, PhD (Other)
Collaborators: EMD Serono (Industry); The Applebaum Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Panagiotis Konstantinopoulos, MD, PhD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-301
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; ARID1A Gene Mutation; Recurrent Endometrial Carcinoma
Keywords: Endometrial Cancer; ARID1A Mutated Recurrent Endometrial Cancer; Recurrent Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and M1774 (Experimental): 25 participants will be enrolled and complete study procedures. The first 6 participants enrolled will take part in a lead-in phase with a dose de-escalation plan for M1744, starting at Dose Level 0 and decreasing to Dose Level -1 and then -2 if applicable per the protocol depending on the occurrence of dose-limiting toxicities. Participants will complete:
  * Baseline visit with assessments and CT or MRI scan.
  * CT or MRI scans every 12 weeks
  * Cycle 1 through End of Treatment:
    * Days 1 - 14 and 22 - 35 of 42-day Cycle: Predetermined dose of M1774 1x daily.
    * Days 1, 15, 29 of 42-day Cycle: Predetermined dose of Avelumab 1x daily.
  * End of Treatment visit with with CT or MRI scan
  * 30 day post-treatment follow up visit
  * 90 day post-treatment follow up
  * Long term follow up every 6 months for up to 3 years.
  Interventions: Drug: Avelumab; Drug: M1774

INTERVENTIONS:
Drug: Avelumab — Human IgG1 antibody, 20mL single-use vials, via intravenous (into the vein) infusion per protocol.
  Other Names: MSB0010718C
Drug: M1774 — Ataxia Telangiectasia and Rad3-related protein (ATR) inhibitor, 30 and 50 mg capsules, taken orally per protocol.
  Other Names: MSC2584415A; Tuvusertib; VXc-400; VRT-1363004; 2-Amino-6-fluoro-pyrazolo[1,5-a] pyrimidine-3-carboxylic acid [5-fluoro-4-(3-methyl-3H-imidazol-4-yl)-pyridin-3-yl]-amide

SUMMARY:
The purpose of this research study is to see if the combination of study drugs avelumab and M1774 is effective and safe for participants with endometrial cancer.

The names of the study drugs involved in this study are:

* Avelumab (a type of human IgG1 antibody)
* M1774 (a type of ATR inhibitor)

DETAILED DESCRIPTION:
This is a non-randomized, open-label, two-stage, phase 2 trial of avelumab in combination with ATR inhibitor (ATRi) M1774 in participants with ARID1A-mutated endometrial cancers who have received prior immunotherapy.

The U.S. Food and Drug Administration (FDA) has not approved avelumab for ARID1A-mutated recurrent endometrial cancer but it has been approved for other uses. The FDA has not approved M1774 as a treatment for any disease.

The research study procedures including screening for eligibility, in-clinic treatment visits, blood tests, urine tests, Computerized Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans, and electrocardiograms (ECGs).

Participants will receive study treatment for up to 2 years and will be followed for up to 3 years until the study is complete.

It is expected that about 25 people will take part in this research study.

EMD Serono is supporting this research study by providing the study drugs avelumab and M1774.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have endometrial cancer that is ARID1A-mutated [loss of function (LOF) mutations] determined by any CLIA-certified next-generation sequencing assay. ARID1A LOF mutation status must be confirmed by the principal investigator prior to participant enrollment.
* Participants must have measurable disease per RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions). Each lesion must be >= 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI.
* Prior Therapy: There is no upper limit of prior therapies, but patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma. Initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy. Furthermore, patients who have only received chemotherapy with immunotherapy in the adjuvant setting will be eligible for the study.

  --Prior hormonal therapy is allowed (no washout period is required after hormonal therapy).
* Participants must have received prior immunotherapy targeting the PD-1/PD-L1 pathway either in the adjuvant, first-line or recurrent setting. Up to 50% of participants (i.e. a maximum of 12 participants) who do not meet this requirement may enroll in the study.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of the combination of avelumab and M1774 in participants <18 years of age, children are excluded from this study.
* ECOG performance status 0, 1, or 2 (reference Appendix A for ECOG performance status criteria).
* Availability of a formalin fixed paraffin embedded (FFPE) block of cancer tissue OR 15 unstained 5-micron slides from the original surgery or biopsy or from a biopsy of recurrent disease.
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Hemoglobin ≥ 9.0 g/dL (with no erythropoietin or red blood cell transfusion within the last 14 days)
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN) in the case of documented Gilbert's syndrome, total bilirubin ≤3 x ULN is allowed
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN in patients with documented hepatic involvement, AST/ALT ≤ 5 x ULN is allowed
  * Creatinine clearance ≥ 60 mL/min as estimated by the Cockcroft-Gault formula or institutional standard method OR
  * Glomerular filtration rate (GFR) ≥ 60 mL/min by measured 24-hour urine collection
* The effects of avelumab and M1774 on the developing human fetus are unknown. For this reason and because these agents are known to be teratogenic, women of child-bearing potential must have a negative serum pregnancy test at screening. Women of child- bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 30 days after last avelumab treatment administration and at least 6 months after last M1774 treatment administration. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

  --Women of child-bearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation or salpingectomy, bilateral oophorectomy, or total hysterectomy) or post-menopausal (defined as ≥ 12 months with no menses without an alternative medical cause)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy, immunotherapy, other investigational therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. There is no required washout period for hormonal therapy.
* Participants whose adverse events due to prior anti-cancer therapy have not recovered to ≤ Grade 1, unless toxicity does not constitute a safety risk and/or is stable on supportive therapy in the opinion of the investigator (e.g., alopecia, sensory neuropathy ≤ Grade 2, etc.)
* Participants who are receiving any other investigational agents.
* Participants with clinically controlled brain metastases, which is defined as individuals with central nervous system metastases that have been treated for, are asymptomatic, and have discontinued corticosteroids for > 14 days or are on a stable or decreasing steroid dose (for the treatment of brain metastases) may be enrolled. Participants with meningeal carcinomatosis are excluded.
* Known prior severe hypersensitivity to avelumab or M1774 or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (≥ Grade 3), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Active and/or uncontrolled infection. The following exceptions apply:

  * Participants with HIV infection are eligible if they are on effective antiretroviral therapy with undetectable viral load within 6 months, provided there is no expected drug-drug interaction
  * Participants with evidence of chronic HBV infection are eligible if the HBV viral load is undetectable on suppressive therapy (if indicated), and if they have ALT, AST, and total bilirubin levels < ULN, and provided there is no expected drug- drug interaction
* Participants with a history of HCV infection are eligible if they have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load, and if they have ALT, AST, and total bilirubin levels < ULN.
* Participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day.
* Current or prior use of immunosuppressive medication within 7 days prior to enrollment with the following exceptions to this exclusion criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* History of prior organ transplantation including allogeneic stem-cell transplantation.
* Severe gastrointestinal conditions such as clinical or radiological evidence of bowel obstruction within 4 weeks prior to study entry, uncontrolled diarrhea in the last 4 weeks prior to enrollment, or history of inflammatory bowel disease.
* Participants with psychiatric conditions (including active or recent [within the past year] suicidal ideation of behavior)/social situations that, in the judgment of the investigator, would make the participant inappropriate for study entry.
* Participants with uncontrolled or poorly controlled arterial hypertension, symptomatic congestive heart failure (≥ New York Heart Association Classification Class III), uncontrolled cardiac arrhythmia, unstable angina pectoris, myocardial infarction or a coronary revascularization procedure, cerebral vascular incident, transient ischemic attack, or any other significant vascular disease within 180 days of study intervention start.
* Known alcohol or drug abuse.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years or if they are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: breast cancer in situ, cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* All other severe acute or chronic medical conditions (for example, immune colitis, inflammatory bowel disease, uncontrolled asthma, immune pneumonitis, or pulmonary fibrosis) or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration in the opinion of the investigator and would make the participant inappropriate for entry into the study.
* Vaccination within 4 weeks of treatment initiation and while on trial is prohibited except for administration of inactivated vaccines.
* Patients may not use natural herbal products or other "folk remedies" while participating in this study. Herbal medications include, but are not limited to St. John's Wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or CYP1A2 enzymes, proton pump inhibitors, or other prohibited concomitant medications within 7 days prior to treatment initiation are ineligible. Examples are provided in Appendix B. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Pregnant women are excluded from this study because avelumab and M1774 are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated with either agent. Women should not breastfeed during the study and for at least 1 month after last treatment administration.
* Calculated QTc average (using the Fridericia correction calculation) of > 470 msec that does not resolve with correction of electrolyte abnormalities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival at 6 months (PFS6) | The observation period related to this endpoint is up to 6 months.
  PFS6 is the percent probability estimate at 6 months based on the Kaplan-Meier method. PFS is defined as the duration of time from study entry to documented disease progression (PD) or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Objective Response Rate (ORR) | The observation period related to this endpoint is up to 2 years.
  ORR was defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) | The observation period related to this endpoint is up to 2 years.
  PFS based on Kaplan-Meier methodology was defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Median Overall Survival (OS) | The observation period related to this endpoint is up to 5 years.
  Overall survival based on the Kaplan-Meier method is defined as the time from registration to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Immune-Related Overall Response Rate(irORR) | The observation period related to this endpoint is up to 2 years.
  irORR was defined as the percentage of participants achieving immune-related complete response (irCR) or immune-related partial response (irPR) on treatment based on irRECIST criteria.
Median Immune-related Progression-free Survival (irPFS) | The observation period related to this endpoint is up to 2 years.
  Immune-related progression-free survival (irPFS) rate is defined as time from treatment assignment to death or to immune-related progression of disease (irPD). Per ir RECIST, irPD was defined as Sum of the diameters (longest for non-nodal lesions, shortest for nodal lesions) of target and new measurable lesions increases >= 20% (compared to nadir), confirmed by a repeat, consecutive observation at least 4 weeks from the date first documented, at the investigator's discretion.
Grade 3-5 Treatment-Related Toxicity Rate | The observation period related to this endpoint is up to 2 years.
  The percentage of participants who experienced a maximum grade 3-5 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv4) as reported on case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu